CLINICAL TRIAL: NCT03005860
Title: A Prospective, Randomized, Controlled Trial to Compare the Effect of TIVA Propofol vs Sevoflurane Anaesthetic on Serumserum Biomarkers and on PBMCs in Patients Undergoing Breast Cancer Resection Surgery
Brief Title: Effect of TIVA Propofol vs Sevoflurane Anaesthetic on Serum Biomarkers and on PBMCs in Breast Cancer Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding could not be arranged, so the study was prematurely terminated
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr. J. V. Divatia, Professor and Head, Department Of Anaesthesia, Critical Care and Pain, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PN 219
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2020-03

CONDITIONS: Female Breast Cancer
MeSH Terms: interventions — Propofol; Sevoflurane; Fentanyl; Atracurium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoromethyl hexafluoroisopropyl ether (Active Comparator): In Sevoflurane group, anaesthesia will be induced with Thiopental 5 - 7mg/kg, fentanyl citrate 2mcg/kg and atracurium besylate 0.5mg /kg to facilitate LMA placement. Anaesthesia will be maintained with sevoflurane 2-2.2 % to maintain a target MAC value between 0.8 & 1.0.
  Interventions: Drug: Fluoromethyl hexafluoroisopropyl ether; Drug: Fentanyl Citrate; Drug: Atracurium Besylate
- 2,6 diisopropylphenol (Experimental): In Propofol group, anesthesia will be will be induced with Propofol TCI [target controlled infusion pump - Injectomat® TIVA Agilia (Fresenius Kabi)] using Schneider model to achieve target site concentration of 4-6mcg/ml, fentanyl citrate 2mcg/kg and atracurium besylate 0.5mg /kg to facilitate LMA placement. Anaesthesia will be maintained with TCI propofol at 3 - 6 mcg/ml as effect site concentration to maintain BIS 40-60.
  Interventions: Drug: 2,6-Diisopropylphenol; Drug: Fentanyl Citrate; Drug: Atracurium Besylate

INTERVENTIONS:
Drug: 2,6-Diisopropylphenol — In Propofol group, anesthesia will be induced with Propofol TCI using Schneider model to achieve a target site concentration of 4 - 6 mcg/ml. Propofol TCI to achieve BIS (Bispectral Index) between 40-60.
  Other Names: Fresofol 1%, Fresenius Kabi
  Arms: 2,6 diisopropylphenol
Drug: Fluoromethyl hexafluoroisopropyl ether — In Sevoflurane group, anesthesia will be induced with 5 - 7mg/kg thiopental, maintenance with O2 with air 50:50%, sevoflurane 2-2.5 %, Further fentanyl, in increments of 1 mcg/kg - and atracurium 0.15 mg/kg, will be given as indicated by the clinical signs and hemodynamic changes.
  Other Names: Sevoflurane
  Arms: Fluoromethyl hexafluoroisopropyl ether
Drug: Fentanyl Citrate — Inj. fentanyl 2 mcg/kg will be used as an adjunct during anaesthetic induction.
  Other Names: Verfen 100mcg/2ml, Verve
Drug: Atracurium Besylate — Inj. atracurium 0.5 mg/kg for will be administered for facilitating LMA placement
  Other Names: Atrapure 25mg/2.5ml, Samarth Life Sciences Pvt. Ltd.

SUMMARY:
Surgery, perioperative stress, anaesthetics and analgesics may modulate the immunosurveillance mechanisms and overwhelm host defences that normally maintain a balance between immunity & carcinogenesis. This may lead to escape of cancer cells and tilt the scales toward a more protumorigenic microenvironment. Volatile agents, in particular, have been shown to exhibit profound immunosuppressive effects. In comparison, propofol has a favorable profile and inhibits cancer cell activity. Determining "cancer-protective" role of TIVA with propofol presents an exciting window of opportunity that has potential to improve outcomes in cancer patients undergoing resection surgery

DETAILED DESCRIPTION:
For the current study, consenting patients planned for upfront surgery, will be randomly allocated to 2 groups- 20 patients each group: Propofol TCI-based Total Intravenous Anesthesia group (Propofol group) and Sevoflurane group (Sevoflurane group), according to computer generated randomization number.

Patients will be monitored routinely with ECG, non invasive blood pressure, and a pulse- oximetery (SPO2), every 5 min. An intravenous access will be established with 20- 22 G cannula. A perioperative antibiotic prophylaxis will be given to all patients. None of the patients will receive any premedication.

After preoxygenation with 100% O2 for 3 min: group specific separate interventions will be performed.

Patient will be ventilated with TV of 6-8ml/kg,respiratory rate will be adjusted to maintain end-tidal CO2 value between 40 - 45 mmHg. Crystalloids will be used for hydration (4-6 ml/kg/h), and intraoperative volume deficits will be replaced by additional administration of a solution according to clinical needs. For TIVA group, the depth of anaesthesia will be monitored using Bispectral Index, with target BIS value between 40 and 60. For Sevoflurane group, the depth of anaesthesia will be monitored using MAC, with target MAC value between 0.8 and 1. Half hour before conclusion of surgery, all patients will receive 0.1mg/kg of ondansetron as prophylaxis for PONV. At the end of surgery, muscle relaxation will be reversed by glycopyrrolate (10mcg/kg) and neostigmine (50mcg/kg).

Patients in both groups will receive intra-venous non-steroidal anti-inflammatory drug 1-1.5mg/kg diclofenac + Paracetamol 1gm just before conclusion of surgery for postoperative analgesia. Postoperative pain & PONV will be managed as per institutional protocols.

ASSAY Peripheral blood (5ml) will be collected from patients in EDTA vaccutainer and (5ml) in another vaccutainer containing clot activator. The sample will be collected at following time points.

1. before anaesthesia (Tpre)
2. after removal of tumor intraoperative (Ti)
3. 2 h after surgery (T2h) , and
4. (T24h) 24 hours after surgery

Estimation of serum cytokines : by sandwich ELISA and by cytokine bead array (CBA) method.

Expression of various lymphocyte subsets (CD3+ T cells, CD4+ helper T cells, CD8+ cytotoxic T cells, γδT cells, NK cells and B cells) by flow cytometry

ELIGIBILITY:
Inclusion Criteria:

1. Women with histopathologically (biopsy/FNAC) proven breast carcinoma with Resectable disease (T 1-4, N 0-1, M 0) [Stage I-III].
2. Willing for upfront modified radical mastectomy.
3. ASA Physical Status 1-2

Exclusion Criteria:

1. use of morphine or on steroid therapy upto 3 months before surgery;
2. history of substance abuse or cognitive dysfunction;
3. endocrine disorders- diabetes, hypothyroid;
4. history of HIV, Hep-B or Hep-C infections;
5. Contraindication to analgesics or anaesthetic drugs;
6. Pregnant & lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline levels versus 24 hour postoperative levels (Tpre vs T24h ) of serum HIF-1a and VEGF-C in both groups. | Baseline levels versus 24 hour postoperative levels (Tpre vs T24h )
  The primary objective of this study is to compare the potential effects of inhalation anesthetic (Sevoflurane) with intravenous anesthetic agent (Propofol) on preoperative levels versus 24hour postoperative levels (Tpre vs T24h ) of serum Hypoxia Inducible Factor-1 alpha (HIF-1a) and Vascular Endothelial Growth Factor -C (VEGF-C) in patients with breast cancer undergoing resection surgery.

SECONDARY OUTCOMES:
Change in levels of serum biomarkers HIF-1a & VEGF-C in patients with breast cancer undergoing resection surgery at other time points - intraoperative, at 2hr postoperative. Ti, T2h in both groups. | after removal of tumor intraoperative (Ti) and 24 hours after surgery (T24h)
  Change in levels of serum biomarkers HIF-1a & VEGF-C in patients with breast cancer undergoing resection surgery at other time points - intraoperative, at 2hr postoperative. Ti, T2h in both groups
Change in levels of serum biomarkers TGF-β, IL-17 IFN-g, TNF-a, IL-6 and MMP-2 at the four time points in both groups. | preoperative, intraoperative, at 2hr postoperative and at 24hr postoperative.
  Transforming Growth Factor -beta (TGF-β), Interleukin - 17 (IL-17), Inferferon - gamma (IFN-g), Tumor Necrosis Factor - alpha (TNF-a), Interleukin - 6 (IL-6), Matrix Metalloproteinase - 2 (MMP-2)
Measure expression of various lymphocyte subsets (CD3+ T cells, CD4+ helper T cells, CD8+ cytotoxic T cells, γδT cells, NK cells and B cells peripheral blood lymphocytes at four time points | preoperative, intraoperative, at 2hr postoperative and at 24hr postoperative.
  Measure expression of various lymphocyte

CONTACTS AND LOCATIONS:
Overall Officials: Shubhada Chiplunkar, Study Chair — Tata Memorial Centre; Rajan Badwe, Study Chair — Tata Memorial Centre; Anuja Bidkar, Study Chair — Tata Memorial Centre; Reshma Ambulkar, Study Chair — Tata Memorial Centre; Raghu Thota, Study Chair — Tata Memorial Centre; Vani Parmar, Study Chair — Tata Memorial Centre
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dikshit RP, Yeole BB, Nagrani R, Dhillon P, Badwe R, Bray F. Increase in breast cancer incidence among older women in Mumbai: 30-year trends and predictions to 2025. Cancer Epidemiol. 2012 Aug;36(4):e215-20. doi: 10.1016/j.canep.2012.03.009. Epub 2012 Apr 20. PMID 22521561
- [Result] Weigelt B, Peterse JL, van 't Veer LJ. Breast cancer metastasis: markers and models. Nat Rev Cancer. 2005 Aug;5(8):591-602. doi: 10.1038/nrc1670. PMID 16056258
- [Result] Dunn GP, Old LJ, Schreiber RD. The immunobiology of cancer immunosurveillance and immunoediting. Immunity. 2004 Aug;21(2):137-48. doi: 10.1016/j.immuni.2004.07.017. PMID 15308095
- [Result] Tavare AN, Perry NJ, Benzonana LL, Takata M, Ma D. Cancer recurrence after surgery: direct and indirect effects of anesthetic agents. Int J Cancer. 2012 Mar 15;130(6):1237-50. doi: 10.1002/ijc.26448. Epub 2011 Nov 9. PMID 21935924
- [Result] Tsuchiya Y, Sawada S, Yoshioka I, Ohashi Y, Matsuo M, Harimaya Y, Tsukada K, Saiki I. Increased surgical stress promotes tumor metastasis. Surgery. 2003 May;133(5):547-55. doi: 10.1067/msy.2003.141. PMID 12773983
- [Result] Boomsma MF, Garssen B, Slot E, Berbee M, Berkhof J, Meezenbroek Ede J, Slieker W, Visser A, Meijer S, Beelen RH. Breast cancer surgery-induced immunomodulation. J Surg Oncol. 2010 Nov 1;102(6):640-8. doi: 10.1002/jso.21662. PMID 20677220
- [Result] Camara O, Kavallaris A, Noschel H, Rengsberger M, Jorke C, Pachmann K. Seeding of epithelial cells into circulation during surgery for breast cancer: the fate of malignant and benign mobilized cells. World J Surg Oncol. 2006 Sep 26;4:67. doi: 10.1186/1477-7819-4-67. PMID 17002789
- [Result] Divatia JV, Ambulkar R. Anesthesia and cancer recurrence: What is the evidence? J Anaesthesiol Clin Pharmacol. 2014 Apr;30(2):147-50. doi: 10.4103/0970-9185.129990. No abstract available. PMID 24803747
- [Result] Heaney A, Buggy DJ. Can anaesthetic and analgesic techniques affect cancer recurrence or metastasis? Br J Anaesth. 2012 Dec;109 Suppl 1:i17-i28. doi: 10.1093/bja/aes421. PMID 23242747
- [Result] Melamed R, Bar-Yosef S, Shakhar G, Shakhar K, Ben-Eliyahu S. Suppression of natural killer cell activity and promotion of tumor metastasis by ketamine, thiopental, and halothane, but not by propofol: mediating mechanisms and prophylactic measures. Anesth Analg. 2003 Nov;97(5):1331-1339. doi: 10.1213/01.ANE.0000082995.44040.07. PMID 14570648
- [Result] Mammoto T, Mukai M, Mammoto A, Yamanaka Y, Hayashi Y, Mashimo T, Kishi Y, Nakamura H. Intravenous anesthetic, propofol inhibits invasion of cancer cells. Cancer Lett. 2002 Oct 28;184(2):165-70. doi: 10.1016/s0304-3835(02)00210-0. PMID 12127688
- [Result] Looney M, Doran P, Buggy DJ. Effect of anesthetic technique on serum vascular endothelial growth factor C and transforming growth factor beta in women undergoing anesthesia and surgery for breast cancer. Anesthesiology. 2010 Nov;113(5):1118-25. doi: 10.1097/ALN.0b013e3181f79a69. PMID 20930611
- [Result] Xu YJ, Chen WK, Zhu Y, Wang SL, Miao CH. Effect of thoracic epidural anaesthesia on serum vascular endothelial growth factor C and cytokines in patients undergoing anaesthesia and surgery for colon cancer. Br J Anaesth. 2014 Jul;113 Suppl 1:i49-55. doi: 10.1093/bja/aeu148. Epub 2014 Jun 25. PMID 24966150
- [Result] Wigmore TJ, Mohammed K, Jhanji S. Long-term Survival for Patients Undergoing Volatile versus IV Anesthesia for Cancer Surgery: A Retrospective Analysis. Anesthesiology. 2016 Jan;124(1):69-79. doi: 10.1097/ALN.0000000000000936. PMID 26556730
- [Result] Gisterek I, Matkowski R, Kozlak J, Dus D, Lacko A, Szelachowska J, Kornafel J. Evaluation of prognostic value of VEGF-C and VEGF-D in breast cancer--10 years follow-up analysis. Anticancer Res. 2007 Jul-Aug;27(4C):2797-802. PMID 17695450